CLINICAL TRIAL: NCT03682315
Title: Algae-derived Hydroxyapatite Behaviour as Bone Biomaterial in Comparison to Anorganic Bovine Bone. A Randomised Split-mouth Human Study.
Brief Title: Comparison of Phicogenic vs. Xenogeneic Biomaterial for Maxillary Sinus Floor Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Pablo Galindo-Moreno, Full Professor of Oral Surgery and Implant Dentistry, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 307CEIH2017
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Sinus Floor Augmentation
Keywords: Maxillary sinus augmentation; Sinus lift; Biomaterial; Anorganic bovine bone; Phicogenic biomaterial; Implant Dentistry

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biphasic phycogenic biomaterial (Active Comparator): Biphasic phycogenic biomaterial and Autogenous cortical bone
  Interventions: Device: Biphasic phycogenic biomaterial
- Xenograft bovine hydroxyapatite (Experimental): Xenograft bovine hydroxyapatite and Autogenous cortical bone
  Interventions: Device: Xenograft bovine hydroxyapatite

INTERVENTIONS:
Device: Biphasic phycogenic biomaterial — Maxillary sinus floor elevation and bone grafting with the use of biphasic phycogenic biomaterial combined with autogenous cortical bone
  Arms: Biphasic phycogenic biomaterial
Device: Xenograft bovine hydroxyapatite — Maxillary sinus floor elevation and bone grafting with the use of xenograft bovine hydroxyapatite combined with autogenous cortical bone
  Arms: Xenograft bovine hydroxyapatite

SUMMARY:
The study aims to evaluate the clinical and radiological behavior, the histological and morphometrical components, the expression of proteins related to bone formation, and the analysis of markers of reparative mesenchymal stromal cells, after using a biphasic phicogenic biomaterial in comparison with anorganic bovine bone.

A randomized split-mouth clinical study is designed to include patients in need of two-stage bilateral maxillary sinus floor elevation. Patients are assigned to receive a mix of autogenous bone and a biphasic phycogenic biomaterial in one maxillary sinus and a mix of autogenous bone and xenograft bovine hydroxyapatite in the other maxillary sinus. Cone-beam computerized tomography (CBCT) scans are performed before sinus floor elevation and 6 months after the procedure to assess the bone gain. Bone core biopsies are obtained at the site of implant placement 6 months after the floor elevation. Histological sections are subjected to histomorphometric and immunohistochemical evaluation of differentiation markers.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients.
* Kennedy class I in the upper jaw.
* Less than 5 mm of residual crestal bone to the maxillary sinus.
* Need for the replacement of teeth with dental implants.

Exclusion Criteria:

* Sinus pathology (sinusitis, mucocele, cysts).
* Smokers.
* Previous long-term (>3 months) use of drugs known to affect bone metabolism, such as bisphosphonates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Sinus floor height change | From surgery to 6 months
  CBCT scans are performed before the sinus floor elevation and 6 months later before implant placement to calculate vertical bone height change from the crestal bone to the floor of the maxillary sinus

SECONDARY OUTCOMES:
Area of new mineralized tissue | 6 months
  Histomorphometric quantification of new mineralized tissue in a bone biopsy collected 6 months after the grafting procedure
Area of non-mineralized tissue | 6 months
  Histomorphometric quantification of non-mineralized tissue in a bone biopsy collected 6 months after the grafting procedure
Area of remaining graft particles | 6 months
  Histomorphometric quantification of remaining graft particles in a bone biopsy collected 6 months after the grafting procedure

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Galindo-Moreno, DDS, PhD, MS, Principal Investigator — Universidad de Granada
Locations (1):
- Facultad de Odontología, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galindo-Moreno P, Hernandez-Cortes P, Mesa F, Carranza N, Juodzbalys G, Aguilar M, O'Valle F. Slow resorption of anorganic bovine bone by osteoclasts in maxillary sinus augmentation. Clin Implant Dent Relat Res. 2013 Dec;15(6):858-66. doi: 10.1111/j.1708-8208.2012.00445.x. Epub 2012 Feb 29. PMID 22376122
- [Background] Galindo-Moreno P, Avila G, Fernandez-Barbero JE, Aguilar M, Sanchez-Fernandez E, Cutando A, Wang HL. Evaluation of sinus floor elevation using a composite bone graft mixture. Clin Oral Implants Res. 2007 Jun;18(3):376-82. doi: 10.1111/j.1600-0501.2007.01337.x. Epub 2007 Mar 12. PMID 17355356
- [Background] Galindo-Moreno P, de Buitrago JG, Padial-Molina M, Fernandez-Barbero JE, Ata-Ali J, O Valle F. Histopathological comparison of healing after maxillary sinus augmentation using xenograft mixed with autogenous bone versus allograft mixed with autogenous bone. Clin Oral Implants Res. 2018 Feb;29(2):192-201. doi: 10.1111/clr.13098. Epub 2017 Oct 26. PMID 29071736
- [Result] Galindo-Moreno P, Padial-Molina M, Lopez-Chaichio L, Gutierrez-Garrido L, Martin-Morales N, O'Valle F. Algae-derived hydroxyapatite behavior as bone biomaterial in comparison with anorganic bovine bone: A split-mouth clinical, radiological, and histologic randomized study in humans. Clin Oral Implants Res. 2020 Jun;31(6):536-548. doi: 10.1111/clr.13590. Epub 2020 Mar 6. PMID 32072685